CLINICAL TRIAL: NCT05425979
Title: Onset of Sensory Blockade in Ultrasound-Guided Ankle Block With Mepivacaine Versus Bupivacaine: A Randomized Non-Inferiority Clinical Trial
Brief Title: Mepivacaine Versus Bupivacaine Onset Time in Ultrasound-guided Ankle Blocks
Status: Enrolling by invitation | Phase: Phase 4 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Bridget P. Pulos, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 22-000140
Record Dates: First submitted 2022-06-16; First posted 2022-06-21 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Ankle Block; Foot Surgery
Keywords: Ultrasound-Guided Ankle Block; Regional anesthesia; Local anesthesia
MeSH Terms: interventions — Mepivacaine; Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Participants, the anesthesiologist performing the block and assessing the block efficacy over time will all be masked as to which local anesthetic is being used
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Mepivacaine group (Active Comparator): Subjects will receive an ultrasound-guided peripheral nerve block at the ankle with mepivacaine prior to undergoing foot surgery
  Interventions: Drug: Mepivacaine
- Bupivacaine group (Active Comparator): Subjects will receive an ultrasound-guided peripheral nerve block at the ankle with bupivacaine prior to undergoing foot surgery
  Interventions: Drug: Bupivacaine

INTERVENTIONS:
Drug: Mepivacaine — Up to two 30 ml vials of mepivacaine 1.5% via ultrasound-guided nerve blockade of the tibial and deep peroneal nerves
  Arms: Mepivacaine group
Drug: Bupivacaine — Up to two 30 ml vials of bupivacaine 0.5% via ultrasound-guided nerve blockade of the tibial and deep peroneal nerves
  Arms: Bupivacaine group

SUMMARY:
The purpose of this research is to determine if both local anesthetics (mepivacaine and bupivacaine) are similar in their onset of sensory block to assess the efficiency of ultrasound-guided ankle blocks in our practice. Currently it is the standard of care to perform ankles blocks with both mepivacaine and bupivacaine. However, given similarity in their safety profile researchers would like to compare if one is non-inferior to the other in terms of onset time of ankle block.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 18 years old.
* Patients who provide informed consent to participate.
* Patients undergoing foot surgery who require a peripheral nerve block of the ankle as primary anesthesia.
* ASA (American Society of Anesthesiology) Physical Status Classification I - III.

Exclusion Criteria:

* Inability to consent.
* Allergy to local anesthetic.
* Infection at site of injection.
* Pregnancy.
* Coagulopathy.
* Hepatic or renal failure.
* Preexisting neuropathy in operative limb.
* Planned spinal anesthetic or general anesthesia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-03-11 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-03-30 (Estimated)

PRIMARY OUTCOMES:
Onset of sensory Blockage | 20 minutes
  Time in minutes for successful surgical sensory blockade following the ankle block

SECONDARY OUTCOMES:
Block Failure | 20 minutes
  Number of subjects to experience block failure as defined as opioid administration operatively and /or conversion to general anesthesia
Pain Scores | Post-procedural, approximately 2-4 hours
  Pain scores in post-anesthesia care unit (PACU) will be obtained using the numerical rating scale (0-10 point scale with 0 representing no pain and 10 representing the worst possible pain)
Total opioid received intra-operatively | Intra-operatively, approximately 4-6 hours
  Total amount of opioid received intra-operatively
Time to first opioid use | 24 hours
  Time measured in minutes to the first opioid use
Number of complications | 24 hour
  Total number of procedural complications
Total anesthesia-related time | 20 minutes
  Measured in minutes, defined as performance time plus onset time of local anesthesia
Overall Benefit of Analgesia Score (OBAS) | 24 hours after discharge
  Seven questions to access pain intensity, adverse effects and satisfaction with treatment. Possible score range from 0 to 24, with higher scores indicating worse outcome
Total opioid use after discharge | 24 hours after discharge
  Total amount of opioids used used for pain control after discharge
Duration of the ankle block | 24 hours after discharge
  Length of time measured in minutes the patient to felt until the ankle block completely wore off

CONTACTS AND LOCATIONS:
Overall Officials: Bridget Pulos, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials